CLINICAL TRIAL: NCT03149029
Title: A Phase II Trial of Abbreviated MAPK Targeted Therapy Plus Pembrolizumab in Patients With Unresectable or Metastatic Melanoma
Brief Title: Abbreviated MAPK Targeted Therapy Plus Pembrolizumab in Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ryan J Sullivan, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-642
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BRAFV600 mutant (Experimental): * Pembrolizumab administered intravenously every three weeks
  * Dabrafenib taken every twelve hours orally
  * Trametinib taken every twelve hours orally
  Interventions: Drug: Pembrolizumab; Drug: Dabrafenib; Drug: Trametinib
- BRAFV600 wild type (Experimental): * Pembrolizumab administered intravenously every three weeks
  * Trametinib taken every twelve hours orally
  Interventions: Drug: Pembrolizumab; Drug: Trametinib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a type of antibody that inhibits the cancer cell growth
  Other Names: Keytruda
Drug: Dabrafenib — Dabrafenib is also a cell inhibitor and works by stopping the cancer cell from duplicating
  Other Names: Tafinlar
  Arms: BRAFV600 mutant
Drug: Trametinib — Trametinib is a cell inhibitor that binds to the cancer cells to inhibit the cancer cells' signals to decrease cell growth
  Other Names: Mekinist

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for unresectable or metastatic melanoma.

The drugs involved in this study are:

* Pembrolizumab (Keytruda)
* Trametinib (Mekinist)
* Dabrafenib (Tafinlar)

DETAILED DESCRIPTION:
* This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.
* The FDA (the U.S. Food and Drug Administration) has approved pembrolizumab, dabrafenib, and trametinib for this specific disease but the combination of all three has not been approved.
* This study is being conducted to document whether trametinib with or without dabrafenib taken for brief period of time prior to and with pembrolizumab works better than the investigators expect pembrolizumab to work in participants with unresectable and/or metastatic melanoma. All three of these drugs are FDA-approved for unresectable and/or metastatic melanoma; however, they are not FDA-approved for use all together.

  * Pembrolizumab is a type of antibody that inhibits the cancer cell growth. An antibody is a cell that attaches to other cells to fight off infection.
  * Trametinib is a cell inhibitor that binds to the cancer cells to inhibit the cancer cells' signals to decrease cell growth.
  * Dabrafenib is also a cell inhibitor and works by stopping the cancer cell from duplicating.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed metastatic or unresectable melanoma.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥10 mm with spiral CT scan. See section 11 for the evaluation of measureable disease.
* Participants may have previously received ipilimumab, adjuvant anti-PD1 therapy, or high-dose IL-2. They may not have previously been treated with BRAF inhibitors (vemurafenib, dabrafenib, encorafenib), MEK inhibitors (selumetinib, trametinib, binimetinib, cobimetinib), and/or anti-PD1/PDL1 monoclonal antibodies for metastatic or unresectable disease. Participants must allow 2 weeks between prior chemotherapy targeted small molecule therapy, or radiation therapy prior to study Day 1 or recovery (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of the combination of trametinib with or without dabrafenib, and pembrolizumab in participants less than 18 years of age, children are excluded from this study.
* ECOG performance status ≤1.
* Life expectancy of greater than three months.
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * total bilirubin ≤ 1.5 X institutional upper limits of normal; total bilirubin > 1.5X above institutional upper limits of normal will be allowed if direct bilirubin is within normal limits or if patients has a documented history of Gilbert's disease
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits or creatinine clearance ≥ 60 mL/min/1.73 m2 for subjects with creatinine levels about institutional normal.
* Participants must have BRAFV600-mutation status known.
* Participants must have disease amenable to and be willing to undergo serial core or excisional biopsies of a tumor lesion(s).
* Because both dabrafenib and trametinib are class D agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with either dabrafenib and trametinib, breastfeeding should be discontinued if the mother is treated with either dabrafenib, trametinib, or the combination of dabrafenib and trametinib. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants treated with prior chemotherapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Participants previously treated with BRAF inhibitors (vemurafenib, dabrafenib, encorafenib), MEK inhibitors (selumetinib, trametinib, binimetinib, cobimetinib), and/or anti-PD1/PDL1 monoclonal antibodies for metastatic or unresectable disease. Any other prior therapy will be allowed (including ipilimumab, adjuvant anti-PD1 therapy, high-dose IL-2).
* Participants with symptomatic brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Subjects with asymptomatic, stable brain metastases and/or who have been previously treated for these conditions that are asymptomatic in the absence of corticosteroid therapy are allowed to enroll. Brain metastasis must be stable with verification by imaging (brain MRI completed at screening demonstrating no current evidence of progressive brain metastases.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other anti-neoplastic agents.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Pregnant women are excluded from this study because both dabrafenib and trametinib are class D agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with either dabrafenib and trametinib, breastfeeding should be discontinued if the mother is treated with either dabrafenib, trametinib, or the combination of dabrafenib and trametinib.
* Participants known to be HIV-positive and on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with either dabrafenib or trametinib. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Participants who have had major surgery < 2 weeks prior to entering the study.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* No symptomatic or untreated leptomeningeal disease.
* Participants are not permitted to receive enzyme inducing anti-epileptic drugs.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current/active pneumonitis.
* History of current evidence of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED):
* History of RVO or RPED
* Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or RPED such as evidence of new optic disc cupping, evidence of visual field defects, and intraocular pressure >21 mm Hg.

  * Uncontrolled intercurrent illness including, but not limited to:
  * Ongoing or active infection
  * LVEF <50% as determined by either MUGA scan or Echo
  * Edema > Grade 1
  * Documented myocardial infarction or unstable/uncontrolled cardiac disease (eg, unstable angina, severe arrhythmias, congestive heart failure [New York Heart Association (NYHA) > Class II]) within 6 months of study entry
  * Arterial thrombosis or vascular ischemic events, such as transient ischemic attack, cerebral infarction, within 6 months prior to study entry
  * Serious or non-healing wound
  * History of any medical condition including cardiovascular disease or chronic obstructive pulmonary disease (COPD), that in the opinion of the investigator, may increase the risks associated with study participation or study treatments or may interfere with the conduct of the study or interpretation of study results
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Individuals with a history of a different malignancy are ineligible except for the following circumstances.

  * Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy.
  * Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ and basal cell or squamous cell carcinoma of the skin.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Sullivan, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts general Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 5/14 BRAFV600 mutant patients had clinical benefit and the threshold for opening the BRAFV600 wild type cohort was 9/14 patients. Therefore, no BRAFV600 wild type patients were enrolled.
Groups:
- BRAFV600 mutant: * Pembrolizumab administered intravenously every three weeks
  * Dabrafenib taken every twelve hours orally
  * Trametinib taken every twelve hours orally
  Pembrolizumab: Pembrolizumab is a type of antibody that inhibits the cancer cell growth
  Dabrafenib: Dabrafenib is also a cell inhibitor and works by stopping the cancer cell from duplicating
  Trametinib: Trametinib is a cell inhibitor that binds to the cancer cells to inhibit the cancer cells' signals to decrease cell growth
- BRAFV600 wild type: * Pembrolizumab administered intravenously every three weeks
  * Trametinib taken every twelve hours orally
  Pembrolizumab: Pembrolizumab is a type of antibody that inhibits the cancer cell growth
  Trametinib: Trametinib is a cell inhibitor that binds to the cancer cells to inhibit the cancer cells' signals to decrease cell growth
Period: Overall Study
Arm/Group | BRAFV600 mutant | BRAFV600 wild type
Started | 16 | 0
Completed | 14 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: No BRAFV600 wild type subjects were enrolled due to insufficient funding.
Groups:
- Total: Total of all reporting groups
Arm/Group | BRAFV600 Mutant | BRAFV600 Wild Type | Total
Number analyzed (Participants) | 14 | 0 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (12.4) |  | 58.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 11 |  | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 14 |  | 14
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Clinical Benefit
Description: The rate of clinical benefit is defined as the percentage of patients with stable disease, partial response, or complete response 6 months after the start of treatment per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) while remaining off MAPK-targeted therapy after induction. Response to treatment was assessed using radiographic imaging.
  A partial response (PR) is defined as a decrease in the sum of the longest diameters (SLD) of target lesions greater than or equal to 30%, no new lesions, and no progression of non-target lesions.
  A complete response (CR) is defined as the disappearance of all lesions and pathologic lymph nodes.
  Stable disease is defined as no PR, CR, or progressive disease (PD). PD is defined as an increase in the SLD of target lesions greater than or equal to 20% in comparison with the smallest SLD on study, progression of non-target lesions, or the appearance of new lesions.
Time Frame: 6 months
Population: No BRAFV600 wild type patients were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | BRAFV600 mutant | BRAFV600 wild type
Number analyzed (Participants) | 14 | 0
Participants | 5 |

2. Secondary Outcome: Overall Survival at 1 Year
Description: Overall survival is the time between the first dose of targeted therapy and death from any cause. Overall survival at 1 year is defined as the proportion of participants who were alive one year after starting treatment. For patients who were lost to follow-up or who had no documentation of death at the time of final analysis, follow-up was censored at the date of last assessment of vital status. Confidence intervals are based on log (-log(endpoint)) methodology.
Time Frame: 1 year
Population: No BRAFV600 wild type subjects were enrolled. 2 participants of the original 16 were excluded from the analysis because they didn't receive pembrolizumab, and survival data was not available for 2 additional subjects.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | BRAFV600 mutant | BRAFV600 wild type
Number analyzed (Participants) | 12 | 0
proportion of participants | 0.656 [0.233 to 0.885] |

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the start of study treatment until progressive disease (PD) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) criteria or death due to any cause. Participants alive without disease progression are censored at the the date of last disease evaluation. PD is defined as an increase in the SLD of target lesions greater than or equal to 20% in comparison with the smallest SLD on study, progression of non-target lesions, or the appearance of new lesions. Confidence intervals are based on log (-log(endpoint)) methodology.
Time Frame: Up to 62 months
Population: No BRAFV600 wild type subjects were enrolled. 2 of the original 16 subjects were excluded from the analysis since they didn't receive pembrolizumab, and progression data was not available for one additional subject.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | BRAFV600 mutant | BRAFV600 wild type
Number analyzed (Participants) | 13 | 0
months | 4.73 [3.48 to 6.8] |

ADVERSE EVENTS:
Time Frame: AEs collected up to 2 years, 5 months (from first dose of study treatment until 90 days after the last dose of study treatment.) All cause mortality was assessed up to 62 months.
Description: In addition to the clinicaltrials.gov definitions, (1) Pyrexia accompanied by hypotension, dehydration, renal insufficiency and/or severe (grade 3+) rigors/chills in the absence of an obvious infectious cause, (2) Occurrence of Cutaneous squamous cell carcinoma (SCC), and (3) Central serous retinopathy (CSR) and Retinal Vein Occlusion (RVO) are also considered serious adverse events.
Groups:
- BRAFV600 mutant (Dabrafenib, Trametinib, and Pembrolizumab): * Pembrolizumab administered intravenously every three weeks
  * Dabrafenib taken every twelve hours orally
  * Trametinib taken every twelve hours orally
  Pembrolizumab: Pembrolizumab is a type of antibody that inhibits the cancer cell growth
  Dabrafenib: Dabrafenib is also a cell inhibitor and works by stopping the cancer cell from duplicating
  Trametinib: Trametinib is a cell inhibitor that binds to the cancer cells to inhibit the cancer cells' signals to decrease cell growth
- BRAFV600 mutant (Dabrafenib and Trametinib ONLY): * Dabrafenib taken every twelve hours orally
  * Trametinib taken every twelve hours orally
  Subjects were enrolled to the BRAFV600 mutant arm but did NOT receive pembrolizumab due to toxicity from Dabrafenib/Trametinib and discontinued from the study early. They were therefore excluded from analysis for the primary and secondary outcome measures, but adverse event data is available for these patients.
  Dabrafenib: Dabrafenib is also a cell inhibitor and works by stopping the cancer cell from duplicating
  Trametinib: Trametinib is a cell inhibitor that binds to the cancer cells to inhibit the cancer cells' signals to decrease cell growth
Arm/Group | BRAFV600 mutant (Dabrafenib, Trametinib, and Pembrolizumab) | BRAFV600 wild type | BRAFV600 mutant (Dabrafenib and Trametinib ONLY)
All-Cause Mortality (participants affected / at risk) | 2/14 | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 6/14 | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 13/14 | 0/0 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRAFV600 mutant (Dabrafenib, Trametinib, and Pembrolizumab) (N=14) | BRAFV600 wild type (N=0) | BRAFV600 mutant (Dabrafenib and Trametinib ONLY) (N=2)
Syncope (Nervous system disorders) | 1 (1) | NA | NA
Hypotension (Vascular disorders) | 1 (1) | NA | NA
Sepsis (Infections and infestations) | 1 (1) | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 (1) | NA | NA
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | NA | NA
Rash macro-papular (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
Fever (General disorders) | 2 (4) | NA | NA
Headache (Nervous system disorders) | 1 (1) | NA | NA
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | NA | NA
Diarrhea (Gastrointestinal disorders) | 1 (2) | NA | NA
Dizziness (Nervous system disorders) | 1 (1) | NA | NA
Fatigue (General disorders) | 1 (1) | NA | NA
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | NA | NA
Alanine Aminotransferase Increased (Investigations) | 1 (1) | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRAFV600 mutant (Dabrafenib, Trametinib, and Pembrolizumab) (N=14) | BRAFV600 wild type (N=0) | BRAFV600 mutant (Dabrafenib and Trametinib ONLY) (N=2)
Abdominal Pain (Gastrointestinal disorders) | 6 (12) | NA | 1 (1)
Acne Vulgaris (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | NA | 0
Acute Posterior Vitreous Detachment (Eye disorders) | 1 (1) | NA | 0
Adenoma in Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | 0
Adnexal Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | 0
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | NA | 0
Alanine aminotransferase increased (Investigations) | 3 (10) | NA | 1 (1)
Alkaline phosphatase increased (Investigations) | 4 (11) | NA | 0
Anemia (Blood and lymphatic system disorders) | 5 (9) | NA | 0
Angioma Myolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | 0
Anorexia (Metabolism and nutrition disorders) | 10 (16) | NA | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | NA | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (8) | NA | 0
Aspartate aminotransferase increased (Investigations) | 4 (13) | NA | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | NA | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | NA | 0
Bladder Trabeculation (Hepatobiliary disorders) | 1 (1) | NA | 0
Bloating (Gastrointestinal disorders) | 3 (3) | NA | 0
Blood bilirubin increased (Investigations) | 1 (2) | NA | 0
Blurred vision (Eye disorders) | 2 (5) | NA | 0
Bronchial thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0
Bruising (Injury, poisoning and procedural complications) | 3 (4) | NA | 1 (1)
Cat Bite (Injury, poisoning and procedural complications) | 1 (1) | NA | 0
Chest pain - cardiac (Cardiac disorders) | 1 (2) | NA | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | NA | 0
Chills (General disorders) | 11 (30) | NA | 1 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1) | NA | 0
Cholesterol high (Investigations) | 1 (1) | NA | 0
Cold sore (Infections and infestations) | 1 (1) | NA | 0
Colitis (Gastrointestinal disorders) | 2 (2) | NA | 0
Confusion (Psychiatric disorders) | 1 (1) | NA | 0
Constipation (Gastrointestinal disorders) | 2 (2) | NA | 1 (1)
Cotton wool spots (Eye disorders) | 1 (1) | NA | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | NA | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (9) | NA | 0
Depression (Psychiatric disorders) | 1 (1) | NA | 0
Diaphoresis (General disorders) | 1 (1) | NA | 0
Diarrhea (Gastrointestinal disorders) | 9 (24) | NA | 1 (1)
Diverticulosis (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Dizziness (Nervous system disorders) | 6 (12) | NA | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | NA | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | NA | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (3) | NA | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | NA | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | NA | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | NA | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | NA | 0 (0)
Ear pressure (Ear and labyrinth disorders) | 1 (1) | NA | 0 (0)
Edema limbs (General disorders) | 3 (9) | NA | 0 (0)
Elevated Crp (Blood and lymphatic system disorders) | 1 (1) | NA | 0 (0)
Elevated Lfts (Investigations) | 0 (0) | NA | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 2 (2) | NA | 0 (0)
Erythematous rash (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Esophageal Candidiasis (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (2) | NA | 0 (0)
Eustachian Tube Dysfunction (Ear and labyrinth disorders) | 1 (1) | NA | 0 (0)
Eye pain (Eye disorders) | 2 (2) | NA | 0 (0)
Facial Pain (General disorders) | 1 (2) | NA | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | NA | 0 (0)
Fatigue (General disorders) | 11 (21) | NA | 1 (2)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Fever (General disorders) | 11 (40) | NA | 1 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (3) | NA | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | NA | 0 (0)
Flushing (Vascular disorders) | 1 (3) | NA | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | NA | 0 (0)
Gait disturbance (General disorders) | 2 (2) | NA | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (4) | NA | 0 (0)
Gastrointestinal Disorders - Other: Oral Lesions (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 (0)
GGT increased (Investigations) | 1 (1) | NA | 0 (0)
Headache (Nervous system disorders) | 8 (21) | NA | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | NA | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | NA | 0 (0)
High Frequency Sensorineural Hearing Loss (Ear and labyrinth disorders) | 1 (1) | NA | 0 (0)
Hot flashes (Vascular disorders) | 4 (5) | NA | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (7) | NA | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | NA | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (5) | NA | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | NA | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | NA | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | NA | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | NA | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 6 (13) | NA | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (12) | NA | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | NA | 0 (0)
Hypotension (Vascular disorders) | 4 (6) | NA | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | NA | 0 (0)
Intermittent Lightheadedness (Nervous system disorders) | 1 (1) | NA | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | NA | 0 (0)
Irritability (General disorders) | 1 (1) | NA | 0 (0)
Lamella Macular Hole (Eye disorders) | 1 (1) | NA | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Localized edema (General disorders) | 1 (1) | NA | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | NA | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | NA | 0 (0)
Malaise (General disorders) | 5 (5) | NA | 0 (0)
Mild paraseptal emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 (0)
Musculoskeletal And Connective Tissue Disorders-Other: Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | NA | 0 (0)
Nabothian Cystan (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | 0 (0)
Nail thinning (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | NA | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (15) | NA | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | NA | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | NA | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | NA | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | NA | 0 (0)
Ocular migraine (Eye disorders) | 1 (1) | NA | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (2) | NA | 0 (0)
Pain (General disorders) | 3 (3) | NA | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | NA | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | NA | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | NA | 0 (0)
Papilledema (Eye disorders) | 1 (1) | NA | 0 (0)
Paresthesia (Nervous system disorders) | 3 (4) | NA | 0 (0)
Pigmented bladder nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | NA | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (2) | NA | 0 (0)
Posterior Capsule Opacification (Eye disorders) | 1 (1) | NA | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0 (0)
Pressure with urination (Renal and urinary disorders) | 1 (1) | NA | 0 (0)
Presyncope (Nervous system disorders) | 2 (3) | NA | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | NA | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 6 (8) | NA | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | NA | 0 (0)
Rash macro-papular (Skin and subcutaneous tissue disorders) | 7 (18) | NA | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | NA | 0 (0)
Reproductive System And Breast Disorders-Other: Prostatic Hypertrophy (Reproductive system and breast disorders) | 1 (1) | NA | 0 (0)
Right Ovarian Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | 0 (0)
Seborrheic Keratosis (Skin and subcutaneous tissue disorders) | 3 (3) | NA | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 2 (4) | NA | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | NA | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | NA | 0 (0)
Skin And Subcutaneous Tissue Disorders- Other: Vulvar Lesions (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Skin infection (Infections and infestations) | 1 (3) | NA | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA | 0 (0)
Soreness at site of mass resection (Surgical and medical procedures) | 1 (1) | NA | 0 (0)
Subcutaneous Mass (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | NA | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | NA | 0 (0)
Tenderness at site of biopsy (General disorders) | 1 (1) | NA | 0 (0)
Tenderness left elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Transaminitis (Hepatobiliary disorders) | 1 (1) | NA | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | NA | 0 (0)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | NA | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | NA | 0 (0)
Urinary frequency (Renal and urinary disorders) | 5 (6) | NA | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | NA | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | NA | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (3) | NA | 0 (0)
Urine discoloration (Renal and urinary disorders) | 2 (2) | NA | 0 (0)
Uveitis (Eye disorders) | 1 (1) | NA | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | NA | 0 (0)
Varicose veins (Blood and lymphatic system disorders) | 1 (1) | NA | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | NA | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | NA | 0 (0)
Venous statis changes (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Visual disturbance (Eye disorders) | 1 (1) | NA | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (11) | NA | 0 (0)
Weight loss (Investigations) | 5 (8) | NA | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (4) | NA | 0 (0)
White blood cell decreased (Investigations) | 4 (7) | NA | 0 (0)
Wound infection (Infections and infestations) | 1 (2) | NA | 0 (0)
Xerosis (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)

LIMITATIONS AND CAVEATS:
Only 5/14 BRAFV600 mutant patients had clinical benefit and the threshold for opening the BRAFV600 wild type cohort was 9/14 patients. Therefore, no BRAFV600 wild type patients were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT03149029/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03149029/ICF_001.pdf